CLINICAL TRIAL: NCT02442817
Title: Linagliptin and Mesenchymal Stem Cells: A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Collaborators: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LING-1
Record Dates: First submitted 2015-05-08; First posted 2015-05-13 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Schizophrenia
Keywords: DPP-4 Inhibitor; Linagliptin; SDF1-α
MeSH Terms: conditions — Schizophrenia | interventions — Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Linagliptin patients with schizophrenia (Active Comparator): This group will be made up of 8 participants with schizophrenia and minimal thought disorder who have been stable and taking their prescribed antipsychotics; they will have 12 weeks of treatment and week for assessment. They will receive linagliptin, 5 mg by mouth once per day, while continuing their antipsychotic treatment.
  Interventions: Drug: Linagliptin
- Linagliptin control group (Active Comparator): This group will be made up of 10 control participants with no diagnosis of mental disorder; they will have 12 weeks of treatment and week for assessment. They will receive linagliptin, 5 mg by mouth once per day.
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Linagliptin — 12 weeks of treatment and week for assessment. Linagliptin, 5 mg by mouth once per day for 12 weeks, in combination with continued antipsychotic treatment.
  Other Names: Tradjenta

SUMMARY:
The purpose of the present study is to gather pilot data on the effects of linagliptin on the concentration of the long and short forms of SDF1-α (stromal cell-derived factor alpha) in humans, and to demonstrate the feasibility of such a study in patients with psychosis in our setting.

DETAILED DESCRIPTION:
This study is a 13-week, open-label study of 8 participants with schizophrenia and minimal thought disorder; they will have 12 weeks of treatment and week for assessment. They will receive linagliptin, 5 mg by mouth once per day, while continuing their antipsychotic treatment. The principal outcome measures will be the concentrations of the long and short forms of SDF1-α (stromal cell-derived factor alpha) in blood.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM (Diagnostic and Statistical Manual) criteria for schizophrenia.
* Considered clinically stable, and on the same dose of antipsychotic for two weeks.
* A score no greater than 3 on the PANSS (Positive and Negative Syndrome Scale) Conceptual Disorganization item.
* Not taking any medications for diabetes, or any anti-inflammatories other than occasional aspirin or acetaminophen. Not taking Clozapine.
* Age 18-45 years.
* Can be available for regular morning appointments from 8:00 am to 10:00 am, preferably on Tuesdays, Wednesdays and Thursdays.

Exclusion Criteria:

* Does not meet DSM criteria for substance abuse or dependence.
* No serious current general medical condition, such as cancer, history of stroke or myocardial infarction, tuberculosis, HIV/AIDS, hemophilia, etc.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
SDF1-α (stromal cell-derived factor alpha) Concentration | Blood will be collected on the first week and then biweekly for 12 weeks.

SECONDARY OUTCOMES:
DPP-4 (Dipeptidyl peptidase-4) Activity | Blood will be collected on the first week and then biweekly for 12 weeks.
Monocyte State | Blood will be collected on the first week and then biweekly for 12 weeks.
  Flow cytometry will be used to examine the state of monocytes to look for cells recently arrived from the bone marrow and to examine the polarization (pro-inflammatory vs. anti-inflammatory) of the monocytes
Absolute/Differential leukocyte count | Blood will be collected on the first week and then biweekly for 12 weeks.
  Flow cytometry will be used.
CD271+ cells | Blood will be collected on the first week and then biweekly for 12 weeks.
  Flow cytometry will be used to detect CD271+ cells.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kirkpatrick, MD, Principal Investigator — University of Nevada School of Medicine
Locations (1):
- University of Nevada School of Medicine, Reno, Nevada, United States